CLINICAL TRIAL: NCT03379922
Title: A Randomised Control Trial of Strategies to Maximise Patient Comfort During Extracorporeal Shockwave Lithotripsy
Brief Title: Strategies to Maximise Patient Comfort During ESWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliodhna Browne (Other)
Responsible Party: Sponsor-Investigator, Cliodhna Browne, Specialist Registrar, University College Hospital Galway
Organization: University College Hospital Galway (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCHGESWL
Record Dates: First submitted 2017-12-12; First posted 2017-12-20 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stress balls (Experimental): The first arm will be given stress balls to squeeze during their treatment and will also receive standard care (the offer of oral analgesia)
  Interventions: Behavioral: Stress balls
- Headphones (Experimental): The second arm will be given headphones to listen to music during their treatment and will also receive standard care.
  Interventions: Behavioral: Headphones
- Control (No Intervention): The control group will receive standard care (the offer of oral analgesia)

INTERVENTIONS:
Behavioral: Stress balls — Squeezing stress balls while receiving ESWL treatment
  Arms: Stress balls
Behavioral: Headphones — Listening to music while receiving ESWL treatment
  Arms: Headphones

SUMMARY:
Extracorporeal shockwave lithotripsy is an outpatient treatment for patients with intrarenal calculi. Standard of care involves offering oral analgesia prior to commencing the treatment. Most patients do not take the offered analgesia after the initial treatment. It has been suggested that distraction techniques may be equivalent to oral analgesia in improving tolerability of extracorporeal shockwave lithotripsy treatment. The use of distraction techniques also removes the potential side effects of mediation administration.

DETAILED DESCRIPTION:
The investigators are aiming to assess if distraction techniques help improve patient comfort while undergoing extracorporeal shockwave lithotripsy treatment for renal calculi. Improved tolerability of treatment would result in longer duration of time on the lithotripsy machine and may lead to better stone fragmentation. Outcomes will be completion of treatment and scores on the short form McGill pain questionnaire.

Patients will be randomised into three groups. The randomisation will not be blinded as this is not possible within the design of the study. The first group will be given stress balls to squeeze during treatment and will also receive standard care (the offer of oral analgesia). The second group will be given headphones to listen to music during treatment and will also receive standard care. The third group will receive standard care.

Prior to commencing extracorporeal shockwave lithotripsy, patients will be given the shortened Health Anxiety Inventory score to complete. Following lithotripsy treatment, patients will be given the short form McGill pain questionnaire to complete.

The initial pilot study will aim to recruit sixty patients and further recruitment will take place on the basis of the outcomes of the pilot study.

Inclusion criteria All patients over eighteen years old undergoing extracorporeal shockwave lithotripsy for the first time

Exclusion criteria Patients not capable of giving informed consent Patients in whom extracorporeal shockwave lithotripsy is contraindicated

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* First ESWL treatment

Exclusion Criteria:

* Patients not capable of giving informed consent
* Patients unsuitable for ESWL

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Pain score | At the time of completing lithotripsy treatment (3000 shocks over 40 to 60 minutes)
  Patients will complete the short form McGill pain questionnaire, subdivided into 11 sensory descriptors, 4 affective descriptors and a visual analogue score. Sensory and affective descriptors are each rated as 0-3. Sensory minimum score 0/33 (no pain), maximum score 33/33 (maximum pain). Affective minimum score 0/12 (no pain), maximum score 12/12 (maximum pain). Visual analogue score 0 to 10 (0 being no pain and 10 being worst possible pain).

SECONDARY OUTCOMES:
Early cessation of lithotripsy treatment | At the time of completing lithotripsy treatment (3000 shocks over 40 to 60 minutes)
  Cessation of lithotripsy treatment before completion (3000 shocks over 40-60 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Cliodhna Browne, MRCSI, Principal Investigator — University College Hospital Galway, Ireland
Locations (1):
- University College Hospital Galway, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Browne C, Redmond E, Kelly T, Rogers E, O'Malley P, Nusrat N, Jaffry S, Durkan G, Walsh K, Dowling C, D'Arcy FT. Strategies to maximise patient comfort during extracorporeal shockwave lithotripsy - A randomised controlled trial. Surgeon. 2021 Aug;19(4):207-211. doi: 10.1016/j.surge.2020.07.002. Epub 2020 Aug 6. PMID 32771299